CLINICAL TRIAL: NCT02377414
Title: A Phase I, Subject and Investigator Blind Randomized, Study to Investigate the Pharmacokinetics, Safety and Tolerability of Retosiban in Healthy Japanese Women
Brief Title: Study to Investigate the Pharmacokinetics (PK), Safety and Tolerability of Retosiban in Healthy Japanese Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 117168
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Obstetric Labour, Premature
Keywords: Preterm labor; Retosiban; Pharmacokinetics; Safety; Infusion; GSK2847065
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Retosiban/placebo (Experimental): Each subject in cohort 1 will receive an intravenous (IV) bolus infusion of 6 milligrams (mg) retosiban or placebo over 5 minutes, followed by a continuous infusion of 6 milligram per hour (mg/h) retosiban or placebo for 24 h. At 24 h of dosing, an additional 6 mg retosiban or placebo will be administered over 5 minutes followed by a 12 mg/h infusion over the next 24 h, for a total time of infusion of 48 h. Subjects administered with placebo will receive an equal volume of normal saline as an IV bolus as well as an equal rate of continuous infusion of normal saline as of retosiban.
  Interventions: Drug: Retosiban solution for Infusion; Drug: Placebo
- Cohort 2: Retosiban (Experimental): Each subject in cohort 2 will receive a bolus infusion of 6 mg retosiban over 5 minutes, followed by a continuous infusion of 6 mg/h retosiban for 24 h. At 24 h of dosing, an additional 6 mg retosiban will be administered over 5 minutes followed by a 12 mg/h infusion over the next 24 h, for a total time of infusion of 48 h.
  Interventions: Drug: Retosiban solution for Infusion

INTERVENTIONS:
Drug: Retosiban solution for Infusion — Retosiban will be supplied as clear, colorless IV solution for infusion in 5 mL vial with a unit dose strength of 15 milligrams per milliliter (mg/mL) (each 5 mL vial contains 75 mg retosiban), dosed at up to 300 mg over 48 h infusion
Drug: Placebo — Placebo will be supplied as a clear, colorless IV solution for infusion with a unit dose strength of 0.9% sodium chloride (NaCl) normal saline
  Arms: Cohort 1: Retosiban/placebo

SUMMARY:
This study in healthy, adult Japanese women will characterize the PK, safety and tolerability of retosiban at the therapeutic doses planned to be evaluated in Phase 3. The PK data will be compared to a sub-set of Caucasian women given the same dose of retosiban. This study has two cohorts, cohort 1 will be a double-blind sponsor-open (subjects and investigator blinded and sponsor unblinded), randomized, continuous 48 hours (h) infusion study in healthy, adult Japanese women of child-bearing potential. Cohort 2 is an open label and continuous retosiban 48 h infusion study in Caucasian, adult, healthy women of child bearing potential. So, the PK can be compared with those of Japanese women. Approximately 32 subjects will be enrolled. In cohort 1, approximately 24 subjects will be enrolled and randomized to retosiban and placebo (2:1 ratio) to have 18 women with 12 active, 6 placebo completed subjects. In Cohort 2, 8 subjects will be enrolled to have 6 competed subjects. The total duration of a subject's involvement in this part is anticipated to be up to 6 weeks (including the 28 day screening period).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are between 20 and 45 years and of age, inclusive at the time of signing the informed consent form.
* Japanese, defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese, and that lifestyle including diet has not changed significantly since leaving Japan. Japanese subjects should also have lived outside Japan for less than 10 years.
* Caucasian subjects as defined as an individual having four grandparents who are all descendants of the original peoples of Europe.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring obtained at the screening visit.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the medical monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=43 kilograms (kg) and body mass index (BMI) within the range 17-29.9 kilogram per square meter (kg/m^2) (inclusive).
* Female subjects- A female subject is eligible to participate if she is: A female of non-productive potential secondary to a personal history of a hysterectomy or tubal sterilization procedure.

A female of reproductive potential who is not pregnant (as confirmed by a negative urine or serum human chorionic gonadotropin [hCG] test), not lactating, and agrees to follow one of the options listed in protocol. Contraception requirement for female subjects from 28 days prior to the first dose of study treatment and until completion of the follow-up visit.

* Capable of giving signed informed consent as described in protocol which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QT duration corrected (QTc) >450 milliseconds (msec) NOTES: The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), QT duration corrected for heart rate by Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read.

The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.

* Subjects must abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements) except occasional usage of acetaminophen, within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of investigational product until completion of the follow-up visit, unless in the opinion of the investigator and GlaxoSmithKline (GSK) medical monitor the medication will not interfere with the study.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >7 drinks. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 milliliter [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* History of drug abuse or dependence within 6 months of the study.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2015-04-17 (Actual); Study Completion 2015-04-17 (Actual)

PRIMARY OUTCOMES:
Composite of PK parameters of retosiban administered by intravenous infusion to healthy adult Japanese and Caucasian women of child-bearing potential: AUC, Cmax, t1/2 and clearance of retosiban | Pre-dose, 0.5 h, 1 h, 2 h, 4 h, 8 h, 12 h, 18 h, 24 h (just before dose increase), 24.5 h, 25 h, 26 h, 28 h, 36 h, 42 h, 48 h, 48.5 h, 49 h, 50 h, 52 h, 54 h, 56 h and 60 h post start of the infusion
  PK parameters will include: area under concentration-time curve (AUC), maximum observed concentration (Cmax), terminal phase half-life (t1/2) and clearance (CL) of retosiban
Composite of PK parameters of retosiban and its major inactive metabolite (GSK2847065) in healthy adult Japanese and Caucasian women of child-bearing potential: AUC, Cmax, t1/2 | Pre-dose, 0.5 h, 1 h, 2 h, 4 h, 8 h, 12 h, 18 h, 24 h (just before dose increase), 24.5 h, 25 h, 26 h, 28 h, 36 h, 42 h, 48 h, 48.5 h, 49 h, 50 h, 52 h, 54 h, 56 h and 60 h post start of the infusion
  AUC, Cmax, t1/2

SECONDARY OUTCOMES:
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | Up to 13 days
  AEs and SAEs will be collected from the start of study treatment until the follow-up contact
Composite of clinical laboratory assessments | Up to 13 days
  Clinical laboratory tests will include hematology, clinical chemistry, urinalysis and additional parameters
Vital sign assessment as a measure of safety | Up to 13 days
  Vital signs will be measured in semi-supine position after 5 minutes rest and will include body temperature, systolic and diastolic blood pressure, pulse rate and respiratory rate
Safety as assessed by electrocardiogram (ECG) | Up to 13 days
  Triplicate 12-lead ECGs will be obtained at each time point during the study
Concomitant medication assessment as a measure of safety | Up to 13 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Glendale, California, United States

REFERENCES:
- See also: Results for study 117168 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117168?search=study&b'search_terms=117168'#rs